CLINICAL TRIAL: NCT05029791
Title: Study of Variations of Immune Infiltrate and Cell Plasticity Markers in Patients With Metastatic Melanoma Under Treatment
Brief Title: Variations of Immune Infiltrate and Cell Plasticity Markers in Treated Metastatic Melanoma Patients
Acronym: COLEMAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0906
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: Melanoma; Immune Infiltrate; Cell plasticity markers
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic melanoma (Other): Patients with stage III or IV melanoma eligible for an immunotherapy or targeted therapy
  Interventions: Other: Tumor biopsy; Other: Blood sample

INTERVENTIONS:
Other: Tumor biopsy — 2 cutaneous tumor biopsies before treatment initiation (D-28 to D-1) and under treatment (Month 1)
Other: Blood sample — 1 EDTA blood sample (8mL) before treatment initiation (D-28 to D-1)

SUMMARY:
COLEMAN is an opened prospective monocentric non-randomized study, initiated by the Hospices Civils de Lyon. Population targeted are patients from 18 years old with stage III or IV metastatic melanoma eligible for a metastatic melanoma treatment administered as part of usual care.

The objective is to study the variations of immune infiltrate and cell plasticity before and under immunotherapy or targeted therapy. Two biopsies are done before and one month after the treatment initiation and one blood sample is done after the treatment initiation.

100 patients will be included and followed during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18
* Female patients must agree to the use of 2 methods of contraception. For man one method of contraception is needed if if his partner is in childbearing age throughout the study and for at least 5 months after last study treatment administration.
* Patients with metastatic stage III or IV melanoma relapse
* Eligible for a melanoma metastatic treatment indicated and administered as part of usual care
* Patients must be willing and able to undergo cutaneous tumor biopsies (except on the face and folds or lymph node) according to the study protocol
* Patient insured or beneficiary of a health insurance plan
* Patient able to provide informed consent and sign approved consent forms to participate in the study
* Patient accepting the conservation of biological samples and their use for clinical research including genetic research

Exclusion Criteria:

* Hematologic tumours under treatment
* Patients with a documented history of autoimmune pathology
* Ocular melanoma
* Persons placed under the safeguard of justice
* Use of immunosuppressants including corticosteroids 4 weeks before the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2031-11-18 (Estimated); Study Completion 2031-11-18 (Estimated)

PRIMARY OUTCOMES:
CD8+ T cells | Month 1 before chemotherapy
  Dosage of CD8+ T cells
CD8+ T cells | Month 1 after chemotherapy
  Dosage of CD8+ T cells
expression of ZEB1 protein | Month 1 before chemotherapy
  Dosage of ZEB 1 protein
expression of ZEB1 protein | Month 1 after chemotherapy
  Dosage of ZEB 1 protein

SECONDARY OUTCOMES:
Clinical response | Week 13
  Partial or complete response as assessed by the clinician
Progression free survival | Week 13
  Time between the date of treatment initiation and the date of first progression
Progression free survival | Every year until 5 years
  Time between the date of treatment initiation and the date of first progression
overall survival | Week 13
  Time between the date of treatment initiation and the patient death
overall survival | Every year until 5 years
  Time between the date of treatment initiation and the patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Service de dermatologie (Bâtiment 1A), Lyon, France

IPD SHARING:
Plan to Share IPD: No